CLINICAL TRIAL: NCT01184690
Title: Prospective Trial Comparing Single-Operator and Dual-Operator Double-balloon Endoscopy in Patients With Small-Bowel Disorders
Brief Title: Single-Operator Versus Dual-Operator Double-balloon Endoscopy in Patients With Small-Bowel Disorders
Acronym: DBE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Jian Shi, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DBE-S vs D
Record Dates: First submitted 2010-08-16; First posted 2010-08-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Small-Bowel Disorders
Keywords: double-balloon endoscopy; diagnostic yield

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-operator DBE (Active Comparator): Single-operator double-balloon endoscopy
  Interventions: Procedure: Single-operator double-balloon endoscopy
- Dual-operator DBE (Active Comparator): Dual-operator double-balloon endoscopy
  Interventions: Procedure: dual-operator double-balloon endoscopy

INTERVENTIONS:
Procedure: Single-operator double-balloon endoscopy — Single-operator double-balloon endoscopy
  Arms: Single-operator DBE
Procedure: dual-operator double-balloon endoscopy — dual-operator double-balloon endoscopy
  Arms: Dual-operator DBE

SUMMARY:
Double-balloon endoscopy (DBE) is a new device that allows diagnosis and treatment throughout the entire small intestine. Although the originally described method requires two operators, the investigators have recently developed a method to perform DBE by a single operator. The investigators here assessed the clinical usefulness of this one-person method in comparison to the conventional two-person DBE.

ELIGIBILITY:
Inclusion Criteria:

1. suspected or known small-bowel disease
2. age: 16-70

Exclusion Criteria:

1. pregnancy
2. coagulation disorders
3. prior surgery of the small bowel and colon

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
completion whether the complete enteroscopy is achieved? | 2 hours
  The completion rate for examination of the entire small intestine
lesion-discovery | 2 hours
  lesion-discovery rate

SECONDARY OUTCOMES:
observation time | 2 hours
Number of Participants with Adverse Events | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Jian Shi, MD, Principal Investigator — Shanghai Changzheng Hospital; Bin Shi, MD, Principal Investigator — Shanghai Changzheng Hospital; Wei-Fen Xie, MD, Study Director — Shanghai Changzheng Hospital
Locations (1):
- Shanghai changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Araki A, Tsuchiya K, Okada E, Suzuki S, Oshima S, Okamoto R, Kanai T, Watanabe M. Single-operator method for double-balloon endoscopy: a pilot study. Endoscopy. 2008 Nov;40(11):936-8. doi: 10.1055/s-2008-1077545. Epub 2008 Sep 25. PMID 18819060
- [Result] Araki A, Tsuchiya K, Okada E, Suzuki S, Oshima S, Yoshioka S, Yoshioka A, Kanai T, Watanabe M. Single-operator double-balloon endoscopy (DBE) is as effective as dual-operator DBE. J Gastroenterol Hepatol. 2009 May;24(5):770-5. doi: 10.1111/j.1440-1746.2009.05787.x. Epub 2009 Feb 12. PMID 19220668